CLINICAL TRIAL: NCT04893291
Title: Sirolimus-coated Balloon Versus Drug-eluting Stent in Native Coronary Vessels
Acronym: TRANSFORM II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Ricerca e Innovazione Cardiovascolare ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRANSFORM II
Record Dates: First submitted 2021-05-13; First posted 2021-05-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis
Keywords: DCB; EES; Optical Coherence Tomography (OCT); Sirolimus; Everolimus; TLF
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Everolimus Eluting Stent (Active Comparator)
  Interventions: Device: Everolimus Eluting Stent
- Magic Touch Sirolimus Coated Balloon (Experimental)
  Interventions: Device: Sirolimus Coated Balloon

INTERVENTIONS:
Device: Everolimus Eluting Stent — Patients assigned to this Arm will have an EES implanted after pre-dilatation, the angiography will be conducted as standard of care
  Arms: Everolimus Eluting Stent
Device: Sirolimus Coated Balloon — Patients assigned to this Arm will be treated with Magic Touch Drug Coated Balloon (DCB) after pre-dilatation, the angiography will be conducted as standard of care
  Arms: Magic Touch Sirolimus Coated Balloon

SUMMARY:
International, multicentric, prospective, investigator-driven, open-label, randomized (1:1) clinical trial to observe and evaluate the efficacy, of Magic Touch Sirolimus Coated Balloon (SCB) compared to one of the gold standard treatment for native vessel disease (everolimus-eluting stent, EES).

DETAILED DESCRIPTION:
The purpose of TRANSFORM II study is to observe and evaluate the efficacy of Magic Touch SCB compared to the gold standard treatment for native vessel disease, namely new-generation everolimus-eluting Drug Eluting Stent (DES). Given the inherent and recognized limitations of stents in native vessels with diameter <3 mm, only patients with coronary vessels up to 3.5 mm of diameter (by visual estimation) will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years;
* all patients with a clinical indication to Percutaneous Coronary Intervention (PCI) (stable coronary artery disease or acute coronary syndromes);
* native coronary artery lesion in a vessel with diameter >2.0 mm and ≦3.5 mm at visual estimation;
* maximum lesion length: 50 mm.
* informed consent to participate in the study.

Exclusion Criteria:

* patients with known (and untreatable) hypersensitivity or contraindication to aspirin, heparin, clopidogrel, prasugrel, ticagrelor, sirolimus or contrast media, which cannot be adequately pre-medicated;
* patients participating in another clinical study;
* subject is a woman who is pregnant or nursing (pregnancy test, either urine or blood test must be performed within 7 days prior to the index procedure in woman of child-bearing potential, and must not commit to initiating a pregnancy for 12 weeks after implantation, using effective contraception);
* creatinine clearance <30 ml/min;
* left ventricular ejection fraction <30%;
* life expectancy <12 months;
* ST-elevation myocardial infarction in the previous 48 hours;
* visible thrombus at lesion site;
* culprit lesion stenosis >99% and/or Thrombolysis In Myocardial Infarction (TIMI) flow <2;
* target lesion/vessel with any of the following characteristics:
* concomitant PCI at the same vessel with any device (vessels are considered: left anterior descending, circumflex or right coronary artery);
* pre-dilatation of the target lesion not performed or not successful (residual stenosis >30%);
* severe calcification of the target vessel, at lesion site but also proximally;
* highly tortuous vessel which could impair device delivery to the lesion site following Investigator's judgement;
* previous stent implantation at target vessel (left anterior descending artery; circumflex artery; right coronary artery);
* bifurcation lesion where side branch treatment is anticipated;
* left main stem stenosis >50%;
* target lesion is in left main stem
* Lesion is located within asaphenous vein graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1820 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of target Lesion Failure (TLF) at 12 Months | 12 Months
  Non-inferiority of Magic Touch SCB compared to everolimus-eluting DES (EES) in terms of target lesion failure (TLF), a composite clinical endpoint, at 12 months.
Number of NACEs | 12 Months
  Verify the superiority of the study device in terms of net adverse clinical events (NACE), a composite endpoint including all-cause death, myocardial infarction (MI), ischemic stroke, and major bleedings following the Bleeding Academic Research Consortium (BARC) types 3 or 5 definition.

SECONDARY OUTCOMES:
Cardiac death | 6, 12, 24, 36, 48 and 60 months
  The occurrence of cardiac death
Death of any cause; | 6, 12, 24, 36, 48 and 60 months
  The occurrence of death of any cause;
Q-wave MI | 6, 12, 24, 36, 48 and 60 months
  The occurrence of Q-wave MI;
MI | 6, 12, 24, 36, 48 and 60 months
  The occurrence of any MI;
Target Lesion Revascularization (TLR) | 6, 12, 24, 36, 48 and 60 months
  The occurrence of TLR;
Target Vessel Revascularization (TVR) | 6, 12, 24, 36, 48 and 60 months
  The occurrence of target vessel revascularization
Bleeding | 6, 12, 24, 36, 48 and 60 months
  The occurrence of bleedings following the BARC classification

CONTACTS AND LOCATIONS:
Locations (53):
- Bangladesh (5):
  - Bangladesh Specialized Hospital Lt, Dhaka
  - Kurmitola General Hospital, Dhaka
  - LABAID Cardiac Hospital, Dhaka
  - National Heart Foundation Hospital & Research Institute, Dhaka
  - National Institute of Cardiovascular Disease, Dhaka
- Brazil (5):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - INC (National Institute of Cardiology),, Rio de Janeiro
  - InCor (Heart Institute), São Paulo
  - Institute Dante Pazzanese of Cardiology, São Paulo
  - Hospital Santa Isabel R. Frei Cornélio, Ubá
- Jurong Park Medical Centre JPMC, Bandar Seri Begawan, Brunei
- France (6):
  - Clinique Louis Pasteur, Essey-lès-Nancy
  - Groupe Hospitalier de La Rochelle, La Rochelle
  - Les Hôpitaux de Chartres, Hôpital Louis Pasteur, Le Coudray
  - Hôpital Prive du Confluent, 4 Rue Éric Tabarly, Nantes
  - Clinique Saint-Hilaire, Rouen
  - Centre Hospitalier de SaintMalo, St-Malo
- Italy (14):
  - Ospedale San Giuseppe Moscati, Aversa
  - Fondazione Poliambulanza, Brescia
  - Ospedale Policlinico San Martino, Genova
  - Ospedale Civile Sant'Andrea, La Spezia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto clinico Sant'Ambrogio, Milan
  - Clinica Polispecialistica San Carlo, Paderno Dugnano
  - A.R.N.A.S. Ospedali Civico Di Cristina Benfratelli, Palermo
  - Azienda Ospedaliera "Ospedali Riuniti Villa Sofia-Cervello", Palermo
  - Ospedale Sandro Pertini, Roma
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma
  - Policlinico Tor Vergata, Roma
  - Ospedale S. Antonio Abate, Trapani
  - Azienda Ospedaliera Universitaria Integrata, Verona
- Malaysia (2):
  - Hospital Queen Elizabeth II, Kota Kinabalu
  - University Malaya Medical Centre (Teaching and Research Hospital), Kuala Lumpur
- Netherlands (5):
  - OLVG Onze Lieve Vrouwe Gasthuis location East, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
  - Erasmus University Medical Center, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Haga Hospital Els Borst, The Hague
- Poland (2):
  - 1st Military Institute of Medicine, Lublin
  - Heliodors Święcicki Clinical Univeristy Hospital, Ul, Poznan
- Spain (8):
  - Hospital General Universitario de Ciudad Real (HGUCR), Ciudad Real
  - Hospital Universitario Lucus Augusti (HULA), Lugo
  - Hospital de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Marqués de Valdecilla (HUMV), Santander
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Alvaro Cunqueiro-University Hospital of Vigo, Vigo
  - Hospital Universitario de Araba, Vitoria-Gasteiz
- Ramathibodi Hospital, Mahidol University, Bangkok, Thailand
- United Kingdom (4):
  - University Hospitals Birmingham, Birmingham
  - Golden Jubilee National Hospital, Clydebank
  - St Bartholomew's Hospital, London
  - Altnagelvin Area Hospital, Londonderry

REFERENCES:
- [Background] Byrne RA, Joner M, Alfonso F, Kastrati A. Drug-coated balloon therapy in coronary and peripheral artery disease. Nat Rev Cardiol. 2014 Jan;11(1):13-23. doi: 10.1038/nrcardio.2013.165. Epub 2013 Nov 5. PMID 24189405
- [Background] Cortese B, Micheli A, Picchi A, Coppolaro A, Bandinelli L, Severi S, Limbruno U. Paclitaxel-coated balloon versus drug-eluting stent during PCI of small coronary vessels, a prospective randomised clinical trial. The PICCOLETO study. Heart. 2010 Aug;96(16):1291-6. doi: 10.1136/hrt.2010.195057. PMID 20659948
- [Background] Cortese B. The PICCOLETO study and beyond. EuroIntervention. 2011 May;7 Suppl K:K53-6. doi: 10.4244/EIJV7SKA9. PMID 22027728
- [Background] Latib A, Colombo A, Castriota F, Micari A, Cremonesi A, De Felice F, Marchese A, Tespili M, Presbitero P, Sgueglia GA, Buffoli F, Tamburino C, Varbella F, Menozzi A. A randomized multicenter study comparing a paclitaxel drug-eluting balloon with a paclitaxel-eluting stent in small coronary vessels: the BELLO (Balloon Elution and Late Loss Optimization) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2473-80. doi: 10.1016/j.jacc.2012.09.020. Epub 2012 Nov 14. PMID 23158530
- [Background] Cortese B, Sgueglia GA, Berti S, Biondi-Zoccai G, Colombo A, Limbruno U, Bedogni F, Cremonesi A; Italian Society of Interventional Cardiology (SICI-GISE). [SICI-GISE position paper on drug-coated balloon use in the coronary district]. G Ital Cardiol (Rome). 2013 Oct;14(10):681-9. doi: 10.1714/1335.14836. Italian. PMID 24121894
- [Background] Cortese B, Berti S, Biondi-Zoccai G, Colombo A, Limbruno U, Bedogni F, Cremonesi A, Silva PL, Sgueglia GA; Italian Society of Interventional Cardiology. Drug-coated balloon treatment of coronary artery disease: a position paper of the Italian Society of Interventional Cardiology. Catheter Cardiovasc Interv. 2014 Feb 15;83(3):427-35. doi: 10.1002/ccd.25149. Epub 2013 Sep 23. PMID 23934956
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] B. Cortese et Al., PICCOLETO II study, JACC Interventions, 2020, in press
- [Background] Scheller B, Vukadinovic D, Jeger R, Rissanen TT, Scholz SS, Byrne R, Kleber FX, Latib A, Clever YP, Ewen S, Bohm M, Yang Y, Lansky A, Mahfoud F. Survival After Coronary Revascularization With Paclitaxel-Coated Balloons. J Am Coll Cardiol. 2020 Mar 10;75(9):1017-1028. doi: 10.1016/j.jacc.2019.11.065. PMID 32138961
- [Background] Lemos PA, Farooq V, Takimura CK, Gutierrez PS, Virmani R, Kolodgie F, Christians U, Kharlamov A, Doshi M, Sojitra P, van Beusekom HM, Serruys PW. Emerging technologies: polymer-free phospholipid encapsulated sirolimus nanocarriers for the controlled release of drug from a stent-plus-balloon or a stand-alone balloon catheter. EuroIntervention. 2013 May 20;9(1):148-56. doi: 10.4244/EIJV9I1A21. PMID 23685303
- [Background] Cortese B, di Palma G, Latini RA, Elwany M, Orrego PS, Seregni RG. Immediate and short-term performance of a novel sirolimus-coated balloon during complex percutaneous coronary interventions. The FAtebenefratelli SIrolimus COated-balloon (FASICO) registry. Cardiovasc Revasc Med. 2017 Oct-Nov;18(7):487-491. doi: 10.1016/j.carrev.2017.03.025. Epub 2017 Mar 25. PMID 28365415
- [Background] Cortese B, Pellegrini D, Latini RA, Di Palma G, Perotto A, Orrego PS. Angiographic performance of a novel sirolimus-coated balloon in native coronary lesions: the FAtebenefratelli SIrolimus COated NATIVES prospective registry. J Cardiovasc Med (Hagerstown). 2019 Jul;20(7):471-476. doi: 10.2459/JCM.0000000000000806. PMID 30994510
- [Background] Cortese B, Testa L, Di Palma G, Heang TM, Bossi I, Nuruddin AA, Ielasi A, Tespili M, Perez IS, Milazzo D, Benincasa S, Latib A, Cacucci M, Caiazzo G, Seresini G, Tomai F, Ocaranza R, Torres A, Perotto A, Bedogni F, Colombo A. Clinical performance of a novel sirolimus-coated balloon in coronary artery disease: EASTBOURNE registry. J Cardiovasc Med (Hagerstown). 2021 Feb 1;22(2):94-100. doi: 10.2459/JCM.0000000000001070. PMID 32740442
- [Background] Kleber FX, Schulz A, Waliszewski M, Hauschild T, Bohm M, Dietz U, Cremers B, Scheller B, Clever YP. Local paclitaxel induces late lumen enlargement in coronary arteries after balloon angioplasty. Clin Res Cardiol. 2015 Mar;104(3):217-25. doi: 10.1007/s00392-014-0775-2. Epub 2014 Oct 28. PMID 25349065
- [Background] Cortese B, Silva Orrego P, Agostoni P, Buccheri D, Piraino D, Andolina G, Seregni RG. Effect of Drug-Coated Balloons in Native Coronary Artery Disease Left With a Dissection. JACC Cardiovasc Interv. 2015 Dec 28;8(15):2003-2009. doi: 10.1016/j.jcin.2015.08.029. Epub 2015 Nov 25. PMID 26627997
- [Background] Onishi T, Onishi Y, Kobayashi I, Sato Y. Late lumen enlargement after drug-coated balloon angioplasty for de novo coronary artery disease. Cardiovasc Interv Ther. 2021 Jul;36(3):311-318. doi: 10.1007/s12928-020-00690-2. Epub 2020 Jul 9. PMID 32647991
- [Derived] Greco A, Sciahbasi A, Abizaid A, Mehran R, Rigattieri S, de la Torre Hernandez JM, Alfonso F, Cortese B. Sirolimus-coated balloon versus everolimus-eluting stent in de novo coronary artery disease: Rationale and design of the TRANSFORM II randomized clinical trial. Catheter Cardiovasc Interv. 2022 Oct;100(4):544-552. doi: 10.1002/ccd.30358. Epub 2022 Sep 2. PMID 36054266